CLINICAL TRIAL: NCT03957291
Title: Chlorohexidine Versus Povidone Iodine as Apreoperative Ophthalmic Disinfectant
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa mohammed mostafa, Asmaa Mohamed Mostafa, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHG vs PI in ophthalmology
Record Dates: First submitted 2019-05-18; First posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Disinfectant Causing Toxic Effect
MeSH Terms: interventions — Chlorhexidine; Povidone-Iodine

STUDY DESIGN:
Intervention Model Description: Randomized prospective trial
Who Masked: Participant
Masking Description: The participant will be masked to which drug they receive, the investigator performing the analysis will also be masked
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Povidine-Iodine (Active Comparator): patients receiving Povidine-Iodine in right eye, chlorhexidine in the left eye before operation
  Interventions: Drug: Povidone-Iodine
- chlorhexidine (Active Comparator): patients receiving Povidine-Iodine in left eye, chlorhexidine in the right eye before operation
  Interventions: Drug: Chlorhexidine

INTERVENTIONS:
Drug: Chlorhexidine — chlorhexidine administration prior to ophthalmic surgery (compared to Povidine iodine )
  Other Names: aqueous Chlorhexidine
  Arms: chlorhexidine
Drug: Povidone-Iodine — Povidine iodine administration prior to ophthalmic surgery (compared to chlorhexidine)
  Other Names: betadine
  Arms: Povidine-Iodine

SUMMARY:
1. Is to assess the efficacy of preoperative disinfection with chlorohexidine and povidone iodine in different concentrations separately .
2. Is to compare the efficacy of chlorohexidine to povidone iodine.
3. Compare patient comfort after instillation of each disinfectant .
4. To find which disinfectant is more effective tolerated and more safe for use .

DETAILED DESCRIPTION:
Methods: This is a single center prospective study comparing antiseptic efficacy and ocular surface irritation with PI (povidine iodine) and AC (aqueous chlorhexidine). . Prior to sugery patients who meet inclusion criteria will be identified and informed consent will be obtained. Study personnel will obtain two samples one from conjunctival sac and th other from skin around the eye. Topical antisepsis will then be applied, the first eye will be randomized to one drop of either PI 5% - 2.5% or AC 0.1%- 0.05% and the second eye will receive the other agent. One minute after instillation of the eye drop to each eye, patients will rate their pain in each eye using the Wong-Baker (smiley face) rating scale. After 15 minutes the second swabs will be taken in the same manner as the first swabs. . On post-operative day three, study personnel will meet the patient and ask to rate the pain in each eye using the same verbal numerical rating scale and to perform slit lamb examination for any complication.

ELIGIBILITY:
Inclusion Criteria:

* Current patient of the Assiute University Hospital arranged for ophthamic surgery
* Age greater than 12.

Exclusion Criteria:

* Documented allergy to PI or AC
* Current diagnosis of infectious keratitis
* History of unilateral contact lens wear in the past 30 days
* Current unilateral use of prescription eye drops.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Patient Comfort | day three post operative
  Patient Comfort using the Wong Baker FACES Pain Scale [Scale: 0(No pain) - 10 (Worst Pain)]

SECONDARY OUTCOMES:
Culture of conjunctiva for bacteria | 7 days
  Microbial flora in conjunctival swab
Patient Comfort | I minute after disinfectant drop instilled
  Patient Comfort using the Wong Baker FACES Pain Scale [Scale: 0(No pain) - 10 (Worst Pain)]

REFERENCES:
- [Background] Grzybowski A, Kanclerz P, Myers WG. The use of povidone-iodine in ophthalmology. Curr Opin Ophthalmol. 2018 Jan;29(1):19-32. doi: 10.1097/ICU.0000000000000437. PMID 28984794